CLINICAL TRIAL: NCT06150703
Title: Luteal Phase Support With GnRH Agonist Alone After GnRH Agonist Triggering and Fresh Embryo Transfer Compared to the Reference Protocol (hCG Triggering and Progesterone Luteal Support): a Randomised Controlled Trial
Brief Title: Luteal Phase Support With GnRH Agonist After GnRH Agonist Triggering in IVF/ICSI Cycles
Acronym: SOLOAGO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220667
Record Dates: First submitted 2023-08-21; First posted 2023-11-29 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: In Vitro Fertilization; ICSI Intracytoplasmic Spermatozoid Injection
Keywords: GnRH agonist triggering; GnRH agonist luteal phase support,; pregnancy; live birth
MeSH Terms: interventions — Ovulation Induction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ovulation triggering with hCG + Luteal phase support with vaginal progesterone (Active Comparator): hCG 250µg subcutaneously between 36h and 38h before oocyte retrieval + Progesterone 600mg/d (200mg tid) vaginally from the evening of the oocyte retrieval until the first pregnancy test
  Interventions: Drug: Ovulation induction with hCG + Luteal phase support with vaginal progesterone
- Ovulation triggering with Triptorelin + Luteal phase support with Nafarelin (Experimental): Triptorelin 0.2 mg subcutaneously between 36h and 38h before oocyte retrieval as a single dose Nafarelin 400µg /day (200µg in the morning 200µg in the evening) nasally from the evening of the oocyte retrieval until the first pregnancy test
  Interventions: Drug: Ovulation triggering by Triptorelin + Luteal phase support by Nafarelin

INTERVENTIONS:
Drug: Ovulation induction with hCG + Luteal phase support with vaginal progesterone — hCG 250µg subcutaneously between 36h and 38h before oocyte retrieval + Progesterone 600mg/d (200mg morning, noon and evening) vaginally from the evening of the puncture until the pregnancy test result
  Arms: Ovulation triggering with hCG + Luteal phase support with vaginal progesterone
Drug: Ovulation triggering by Triptorelin + Luteal phase support by Nafarelin — Triptorelin 0.2 mg subcutaneously between 36h and 38h before oocyte retrieval as a single dose Nafarelin 400µg /day (200µg in the morning 200µg in the evening) nasally from the evening of the oocyte retrieval until the first pregnancy test
  Arms: Ovulation triggering with Triptorelin + Luteal phase support with Nafarelin

SUMMARY:
The development of stimulation protocols for in vitro fertilisation (IVF) has led to a paradox. It has now been established that obtaining a large number of oocytes is a key to success, but that it is also a risk factor for embryo transfer failure after puncture (disruption of endometrial receptivity due to luteal insufficiency) and a risk factor for complications such as ovarian hyperstimulation syndrome (OHSS).

DETAILED DESCRIPTION:
It is currently established that obtaining a large number of oocytes is a key of success in IVF/ICSI cycles. However, it is also a risk factor for ovarian hyperstimulation syndrome (OHSS) and a risk factor of implantation failure after fresh embryo transfer because of the alteration of endometrial receptivity. A freeze all strategy can be proposed to avoid these risks but vitrification of embryos, although more efficient than slow freezing in terms of embryo survival, is not without risk. Furthermore, proper endometrial and embryo timing for frozen-thawed embryo transfer is still debated.

Recent preliminary works suggest another possible way to combine an optimal ovarian response with the recovery of a large number of oocytes, good chances of implantation and a reduced risk of OHSS. To achieve this goal, ovulation triggering and luteal phase support need to be modified together. The human chorionic gonadotropin (hCG) (mimicking the Luteinising Hormone (LH)peak to trigger ovulation) that induces OHSS is replaced by an a GnRH agonist (GnRHa) triggering allowing an endogenous peak of Follicle Stimulating Hormone (FSH) and LH. Then, the usual support of the luteal phase by exogenous vaginal progesterone, whose absorption seems to be suboptimal for about 30% of patients, is replaced by endogenous progesterone production by the corpora lutea, supported by the maintenance of LH activity through the continuation of agonist of gonadotropin releasing hormone (AgoGnRH) in the luteal phase. Pilot studies show that a 10% to 15% increase in ongoing pregnancy rates can be expected with this type of protocol. The objective of our study is to demonstrate an increase in ongoing pregnancy rate per cycle with this new strategy combining GnRHa triggering and GnRHa luteal phase support compared to the reference protocol (hCG triggering and exogenous progesterone luteal phase support).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring conventional IVF or IVF with sperm injection (ICSI) from the partner or donor under the conditions of management defined by French law.
* Patients aged 18 to 39 included
* First or second attempt at IVF or ICSI for pregnancy
* BMI < 35 kg/m2
* Anti-Mullerian hormone (AMH) > 1 ng/ml (= 7 pmol/L) and/or antral follicle count ≥ 8 within the year prior to inclusion
* AMH < 5 ng/ml and/or antral follicle count <40 within the year prior to inclusion
* Treatment with recombinant FSH
* Antagonist protocol (with pre-treatment or not)
* Initial dose of recombinant FSH between 75 and 450 IU
* Signed informed consent
* Affiliation to the social security system (excluding AME)

Exclusion Criteria:

* Patient diagnosed with HIV infection
* ICSI with sperm from testicular biopsy
* Pre-implantation diagnosis
* Hypogonadotropic hypogonadism (amenorrhea or spaniomenorrhea with basal LH <1.2 IU/L)
* History of severe ovarian hyperstimulation syndrome (OHSS)
* Unoperated hydrosalpinx
* Intracavitary polyps or myomas deforming the cavity
* Known hypersensitivity to the investigational drugs and/or their excipients (human chorionic gonadotropin, progesterone, nafarelin acetate, GnRH, GnRH analogues, mannitol, sodium chloride, water for injection, glacial acetic acid, Sodium hydroxide and/or hydrochloric acid, sorbitol, purified water, benzalkonium chloride, sunflower oil, soybean lecithin, gelatin, glycerol, titanium dioxide (E171), methionine, poloxamer 18, phosphoric acid).
* Gynaecological bleeding or genital haemorrhage
* History of epilepsy and/or intracranial tumors potentially causing epilepsy
* Tumours of the hypothalamus or pituitary gland
* Ovarian enlargement or cysts unrelated to polycystic ovary syndrome
* Severe adenomyosis requiring a long protocol
* Carcinoma of the ovary, uterus or breast
* Active thromboembolic events
* Severe impairment of liver function
* Breastfeeding women
* Patients under court protection, guardianship or curators
* Current participation in another therapeutic interventional trial on the day of inclusion
* Patients who do not speak or understand French

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 652 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09-27 (Estimated)

PRIMARY OUTCOMES:
Live birth, defined as the presence of a live birth after 22 weeks' gestation. Twin pregnancies will be counted as a single birth. | 22 weeks' gestation
  To demonstrate an increase in the rate of live births after 22 weeks' amenorrhoea (SA) per cycle with induction and support by GnRH agonist compared with the reference protocol combining induction by hCG and luteal support by exogenous vaginal progesterone

SECONDARY OUTCOMES:
Embryo implantation defined as the presence of a gestational sac on the first ultrasound (5-8 WG) | 5-8 weeks' gestation
  Demonstrate improvement of embryo implantation rates with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Pregnancy defined as an hCG level > 10 IU/ml 14 days after oocyte retrieval. | 14 days after oocyte retrieval.
  Demonstrate an improvement in pregnancy rate with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Clinical pregnancy, defined as an intrauterine gestational sac with embryo showing cardiac activity on ultrasound at 5-10 WG | 5-10 weeks' gestation
  Demonstrate an improvement in clinical pregnancy rate with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Miscarriage prior to 12 WG, defined as the termination of a pregnancy prior to 12 WG. | 12 weeks' gestation
  Demonstrate a decrease in the rate of miscarriage per pregnancy with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Ongoing pregnancy, defined as the presence of an intra-uterine sac with an embryo with cardiac activity visible on ultrasound between 11 weeks of gestations(WG) and 13 WG+6 days (first trimester ultrasound). | first trimester ultrasound (11 weeks of gestation and 13weeks of gestation +6days)
  Demonstrate an increase ongoing pregnancy rate at 12 weeks of gestation (12 WG) per cycle with GnRHa triggering and GnRHa luteal phase support compared with the reference protocol: hCG triggering and exogenous vaginal progesterone luteal phase support.
Number of patients with gravidic hypertension and its onset, | between 12 weeks of gestation and 22 weeks of gestation
  Compare the impact on obstetric data with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Number of patients with pre-eclampsia and its onset, | between 12 weeks of gestation and 22 weeks of gestation
  Compare the impact on obstetric data with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Number of patients with gestational diabetes and its onset | between 12 weeks of gestation and 22 weeks of gestation
  Compare the impact on obstetric data with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Number of patients with term and mode of delivery | between 12 weeks of gestation and 22 weeks of gestation
  Compare the impact on obstetric data with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Number of patients with medical termination of pregnancy | between 12 weeks of gestation and 22 weeks of gestation
  Compare the impact on obstetric data with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Number of patients with late miscarriage (between 12 and 22 WG) | between 12 weeks of gestation and 22 weeks of gestation
  Compare the impact on obstetric data with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Number of patients with fetal death in utero | between 12 weeks of gestation and 22 weeks of gestation
  Compare the impact on obstetric data with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Ovarian hyperstimulation syndrome, defined as the presence of moderate to severe syndrome, early and late. Early defined as the period before D10 post retrieval and late defined as pregnancy related OHSS, after D10 post oocyte retrieval | before Day 10 post retrieval and after Day 10 post oocyte retrieval
  Demonstrate a decrease in the rate of moderate to severe and early and late OHSS with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Progesterone levels on day of oocyte pick up and at Day 7 post oocyte pick up. | Day 7 post oocyte pick up
  Compare the evolution of the corpus luteum in the luteal phase with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Estradiol levels on day of oocyte pick up and at Day 7 post oocyte pick up. | Day 7 post oocyte pick up
  Compare the evolution of the corpus luteum in the luteal phase with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
LH levels on day of oocyte pick up and at Day 7 post oocyte pick up. | Day 7 post oocyte pick up
  Compare the evolution of the corpus luteum in the luteal phase with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
hCG levels on day of oocyte pick up and at Day 7 post oocyte pick up. | Day 7 post oocyte pick up
  Compare the evolution of the corpus luteum in the luteal phase with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Progesterone levels during follow-up, presence of pregnancy and presence of miscarriage. | 19 months
  Assess the association of progesterone levels with pregnancy and miscarriage throughout follow-up with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Estradiol levels during follow-up, presence of pregnancy and presence of miscarriage. | 19 months
  Assess the association of estradiol levels with pregnancy and miscarriage throughout follow-up with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
LH levels during follow-up, presence of pregnancy and presence of miscarriage. | 19 months
  Assess the association of LH levels with pregnancy and miscarriage throughout follow-up with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
hCG levels during follow-up, presence of pregnancy and presence of miscarriage. | 19 months
  Assess the association of hCG levels with pregnancy and miscarriage throughout follow-up with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
All adverse events up to delivery | 19 months
  Evaluate the side effects with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
Number of oocytes collected, | oocyte puncture visit
  Compare embryonic development with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
number of mature oocytes | oocyte puncture visit
  Compare embryonic development with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
number of oocytes fertilised, | 5th day post oocyte puncture visit
  Compare embryonic development with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
number of embryos on the second day of development, | 5th day post oocyte puncture visit
  Compare embryonic development with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
number of blastocysts obtained, | 5th day post oocyte puncture visit
  Compare embryonic development with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
number of blastocysts transferred, | 5th day post oocyte puncture visit
  Compare embryonic development with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.
number of blastocysts frozen. | 5th day post oocyte puncture visit
  Compare embryonic development with GnRHa triggering and GnRHa luteal phase support compared to hCG induction and exogenous vaginal progesterone luteal support.

CONTACTS AND LOCATIONS:
Locations (1):
- Maeliss Peigné, Bondy, France

IPD SHARING:
Plan to Share IPD: No